CLINICAL TRIAL: NCT05432895
Title: Dynamic Versus Static Night Splinting of Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Loretta Chou, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60879
Record Dates: First submitted 2022-05-04; First posted 2022-06-27 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — Splints

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control( static splinting) (Active Comparator): conventional static splint
  Interventions: Device: Dynamic splint
- Experiment( dynamic splinting) (Experimental): Device treats plantar fasciitis and replacing boot immobilization
  Interventions: Device: Dynamic splint

INTERVENTIONS:
Device: Dynamic splint — Device treats plantar fasciitis and replacing boot immobilization which is quite benign

SUMMARY:
The investigators are trying to study that there is no difference in improvement of motion between static progressive and dynamic splinting.

DETAILED DESCRIPTION:
A physical rehabilitation device for the treatment of a medical condition of the foot known as plantar fasciitis includes a splint which is connected to the toe and ankle of a patient. Static splint is the use of inelastic components to apply torque to a joint in order to statically position it as close to end range as possible. A dynamic splint uses a tension spring that is integrated into a brace, usually via a mechanical hinge. The tension spring can be adjusted for more or less tension to achieve range of motion goals with less pain. The investigators are trying to study that there is no difference in improvement of motion between static progressive and dynamic splinting.

ELIGIBILITY:
Inclusion Criteria:

* Demographic - Over 18 years of age and ambulatory without a gait aid with no history of narcotic use
* Diagnosis - Unilateral or bilateral acute (< 6 months of pain) plantar fasciitis (i.e., Heel pain that increases with weightbearing, "First step pain": heel pain that occurs after a period of non-weightbearing, such as in the morning when arising from bed or when arising after prolonged sitting; the pain is improved after a few minutes walking but will worsen again with prolonged weightbearing, tenderness over the medial calcaneal tuberosity at the insertion of the plantar fasciitis)
* Permitted - Icing, NSAIDS( ibuprofen), Custom Shoe Inserts, Diagnostic Ultrasound

Exclusion Criteria:

* Demographic - Under 18 year of age, requires a gait aid for ambulation; if not covered by insurance,
* Diagnosis of - Arthritis of the Ankle, Midfoot, or Forefoot; Inflammatory Arthritis; Gout; Turf Toe; Hallux Rigidus; Hallux Limitus; Sesamoiditis; Tendonitis or Tendinopathy; Prior tear or Rupture of the Plantar Fascia; Fibromyalgia, Neuralgia, or Neuropathy; Peripheral Vascular Disease; Prior Trauma to the Heel, Fracture of the Calcaneus; Infection; Corn; Callus; Ingrown Nail.
* Patient with history of Symptoms for over 6 months
* Refractory to prior splint-based treatments
* Prior injection of the plantar fascia
* Prior surgery on the plantar fascia
* Narcotic use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
NO pain at 1 month follow up | 1 months
  We plan to use VAS pain scale as measurement scale ( range; 0-10, higher scores correspond to greater pain)
NO pain at 3 months follow up | 3 months
  We plan to use VAS pain scale as measurement scale ( range; 0-10, higher scores correspond to greater pain)
NO pain at 6 months follow up | 6 months
  We plan to use VAS pain scale as measurement scale ( range; 0-10, higher scores correspond to greater pain)

SECONDARY OUTCOMES:
Clinically relevant change in Foot Function Index (FFI) | 1 months
  Clinically relevant change in Foot Function Index (FFI) of >6.5 points (MCID
Clinically relevant change in Foot Function Index (FFI) | 3 months
  Clinically relevant change in Foot Function Index (FFI) of >6.5 points (MCID
Clinically relevant change in Foot Function Index (FFI) | 6 months
  Clinically relevant change in Foot Function Index (FFI) of >6.5 points (MCID

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Palo Alto, California
  - Stanford outpatient center, Redwood City, California